CLINICAL TRIAL: NCT02090426
Title: Health Care Hotspotting: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abdul Latif Jameel Poverty Action Lab (Other)
Collaborators: The Cooper Health System (Other); National Bureau of Economic Research, Inc. (Other); Massachusetts Institute of Technology (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JPAL-763
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: High Utilizers of Hospital Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Individuals in the standard care arm receive standard discharge planning from the hospital with no followup by Link2Care team members.
- Link2Care (Experimental): Participants are assigned to a multidisciplinary care team (Link2Care) comprised of a registered nurse, licensed practical nurse, social worker, intervention specialist, community health worker, and health coaches. A representative from the care team engages with the patient at bedside during the hospital admission and plans for the immediate period following discharge. The Program, as a whole, involves a series of home visits, scheduling of and accompaniment to initial primary care and specialty care visits, and support for individuals as they navigate various social service agencies to enroll in public programs including TANF, SNAP, and programs that promote housing stability.
  Interventions: Other: Link2Care

INTERVENTIONS:
Other: Link2Care
  Arms: Link2Care

SUMMARY:
This trial investigates the value created by the highly innovative Camden Coalition of Healthcare Providers' Care Management Program: Link2Care. The program targets "super-utilizers" of the health care system - specifically adults with 2 or more hospitalizations in the last six months 2 or more chronic conditions, and 5 or more outpatient medications - with intensive case management services. In particular, a team of nurses, social workers, community health workers and health coaches, supported by real-time data of healthcare utilization, perform home visits, accompany patients to doctor visits, and help patients enroll in social-service programs. This approach aims to improve the self-sufficiency of patients in navigating the healthcare and social-service systems and has the potential to reduce healthcare costs and improve patient health.

DETAILED DESCRIPTION:
The Camden Coalition of Healthcare Providers' Care Management Program, Link2Care, targets "super-utilizers" of the health care system. These are individuals with medically and socially complex needs who have frequent hospital admissions. Specifically, the Link2Care program targets patients in specific Camden hospitals who have had at least two hospital admissions in the last six months and have at least two chronic conditions.

Such heavy utilizers of hospital care account for a disproportionate share of healthcare spending. For example, CCHP analyzed hospital admission and emergency department use at three Camden hospital systems from 2002-2007 and found that 20% of patients accounted for 90% of the costs (Green et al., 2010). As described below, when we compare patients admitted to Camden hospitals, in the year prior to an admission, a typical patient targeted by the program has 2.5 times more admissions in the prior six months due to the targeting. They are also much more likely to be readmitted to the hospital over the year following the hospital stay, accruing $73,000 in hospital charges over that time compared to $6600 for other patients.

Link2Care provides intensive care management and coordination for up to 6 months following hospital discharge. From October 2012 to January 2014, the median length of the intervention for those who completed it was 85 days.

The approach aims to improve the self-sufficiency of patients in navigating the healthcare and social-service systems. It has the potential to reduce healthcare costs and improve patient health, as patients learn to use primary care to prevent an escalation of symptoms that leads to rehospitalization.

Participants are assigned to a multidisciplinary care team comprised of a registered nurse, licensed practical nurse, social worker, intervention specialist, community health worker, and health coaches. A representative from the care team engages with the patient at bedside during the hospital admission and plans for the immediate period following discharge. Link2Care, as a whole, involves a series of home visits, scheduling of and accompaniment to initial primary care and specialty care visits, and support for individuals as they navigate various social service agencies to enroll in public programs including TANF, SNAP, and programs that promote housing stability.

The patient is enrolled in the program while still in the hospital. Upon discharge, the care team works to visit the patient at home within 3 days of discharge. The care team also works to schedule a primary care visit within 7 days of discharge, and appropriate specialist visits as necessary At the initial home visit, the care team (1) performs medication reconciliation-an inventory of the medications prescribed to gauge appropriateness and patient understanding, (2) conducts an assessment of the patient's perception of the discharge experience and care coordination, medical/health needs, activity/mobility, service needs, and stage of readiness to change, and (3) collaboratively sets goals with the individual, such as compliance with the discharge plan. The care team then works closely with the patient to achieve these goals; as is needed, the team assists the patient in scheduling necessary physician visits, accompanies the patient to those visits, completes applications for social services, and coaches the patient in self-care. Subsequent home visits evaluate the patient's and the team's progress. The end of the intervention is determined based on hospital utilization, individual factors (health education/literacy, disease self-management, skills development, level of engagement, self-efficacy) and some systemic factors (access to, and the quality of, care, social support, etc.). The person receives a graduation certificate. The person is expected to meet their healthcare needs in the future through their primary care physician.

In an earlier, non-randomized evaluation, this program has been found to improve health outcomes, decrease utilization of emergency and inpatient services, and decrease costs for a cohort of 36 "high utilizers" from $1.2 million monthly to $534,000 monthly, a savings of 56% over five years (Green et al., 2010).

Due to staff and financial constraints, Link2Care is currently administered for only a subset of the patients who meet the eligibility criteria, and the patients who are currently approached are chosen in an ad-hoc manner. This study would establish a formal process for determining - via random assignment - which subset of eligible individuals are offered the intervention. This random assignment, which will not reduce the number of individuals who benefit from the services, will allow us to isolate the causal effects of the CCHP Link2Care Program.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following criteria based on the records from the index event:

* Is currently admitted to Cooper or Lourdes hospitals (still in hospital for recruitment)
* Resides in the following zip codes: 08101 (PO zip code), 08102-08105, 08107s, 08110
* Is 19-80 years old
* Has >=2 hospital admissions in the past 6 months (to Camden area hospitals in the Health Information Exchange )
* Has >=2 chronic conditions

Patients must meet at least three of the following criteria based largely on the electronic medical record:

* Has >=5 outpatient medications
* Has difficulty accessing services
* Lacks social support
* Has mental health co-morbidity
* Is actively using drugs
* Is homeless

Exclusion Criteria:

* Already subject in RCT (treatment or control)
* Deceased or discharged prior to triage or recruitment
* Uninsured
* Cognitively impaired
* Oncology patient
* Index hospitalization is for: a surgical procedure for an acute problem, complications of a progressive chronic disease with limited treatments, or mental health issue only with no co-morbid conditions

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy N Finkelstein, PhD, Principal Investigator — The Abdul Latif Jameel Poverty Action Lab/MIT; Jeffery Brenner, MD, Principal Investigator — The Cooper Health System
Locations (2):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - Our Lady of Lourdes Medical Center, Camden, New Jersey

REFERENCES:
- [Derived] Yang Q, Wiest D, Davis AC, Truchil A, Adams JL. Hospital Readmissions by Variation in Engagement in the Health Care Hotspotting Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332715. doi: 10.1001/jamanetworkopen.2023.32715. PMID 37698862
- [Derived] Finkelstein A, Zhou A, Taubman S, Doyle J. Health Care Hotspotting - A Randomized, Controlled Trial. N Engl J Med. 2020 Jan 9;382(2):152-162. doi: 10.1056/NEJMsa1906848. PMID 31914242

RESULTS

PARTICIPANT FLOW:
Groups:
- Link2Care: Participants are assigned to a multidisciplinary care team (Link2Care) comprised of a registered nurse, licensed practical nurse, social worker, intervention specialist, community health worker, and health coaches. A representative from the care team engages with the patient at bedside during the hospital admission and plans for the immediate period following discharge. The Program, as a whole, involves a series of home visits, scheduling of and accompaniment to initial primary care and specialty care visits, and support for individuals as they navigate various social service agencies to enroll in public programs including Temporary Assistance for Needy Families (TANF), Supplemental Nutrition Assistance Program (SNAP), and programs that promote housing stability.
  Link2Care
Period: Overall Study
Arm/Group | Standard Care | Link2Care
Started | 401 | 399
Analysis Population (Subset of randomized participants that matched to discharge data in which we observe outcomes.) | 389 | 393
Completed | 389 | 393
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 12 | 6

BASELINE CHARACTERISTICS:
Population: We report baseline characteristics for the analysis population that matched to hospital discharge data.
Groups:
- Link2Care: Participants are assigned to a multidisciplinary care team (Link2Care) comprised of a registered nurse, licensed practical nurse, social worker, intervention specialist, community health worker, and health coaches. A representative from the care team engages with the patient at bedside during the hospital admission and plans for the immediate period following discharge. The Program, as a whole, involves a series of home visits, scheduling of and accompaniment to initial primary care and specialty care visits, and support for individuals as they navigate various social service agencies to enroll in public programs including TANF, SNAP, and programs that promote housing stability.
  Link2Care
- Total: Total of all reporting groups
Arm/Group | Standard Care | Link2Care | Total
Number analyzed (Participants) | 389 | 393 | 782
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 288 | 279 | 567
  >=65 years | 101 | 114 | 215
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 187 | 391
  Male | 185 | 206 | 391
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 202 | 227 | 429
  Hispanic | 126 | 105 | 231
  Non-Hispanic white | 60 | 58 | 118
  Asian, multiracial, or other | 1 | 3 | 4
Prior Hospital Utilization [Count of Participants; unit: Participants]
  2 admissions in prior year | 165 | 171 | 336
  3+ admissions in prior year | 224 | 222 | 446
Preferred Language [Count of Participants; unit: Participants]
  English | 309 | 329 | 638
  Non-English | 80 | 64 | 144

OUTCOME MEASURES:

1. Primary Outcome: Any Hospital Readmission
Time Frame: 180-day from indexed hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
Participants | 240 | 245

2. Secondary Outcome: Any Emergency Department Use
Time Frame: 180-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

3. Secondary Outcome: Any Hospital Use (Inpatient or ED)
Time Frame: 180-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

4. Secondary Outcome: Inpatient Readmission From the ED
Time Frame: 180-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

5. Secondary Outcome: Inpatient Readmission Not From the ED
Time Frame: 180-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

6. Secondary Outcome: Number of Readmissions
Time Frame: 180-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
readmissions | 1.54 (1.98) | 1.52 (1.98)

7. Secondary Outcome: Had 2+ Readmissions
Time Frame: 180-day from indexed hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
Participants | 141 | 143

8. Secondary Outcome: Number of Days in the Hospital
Time Frame: 180-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: days in hospital
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
days in hospital | 9.95 (14.10) | 9.36 (13.01)

9. Secondary Outcome: Hospital Charges
Time Frame: 180-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: hospital charges ($)
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
hospital charges ($) | 114,768 (187,084) | 116,422 (200,490)

10. Secondary Outcome: Hospital Receipts
Time Frame: 180-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: Hospital Receipts ($)
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
Hospital Receipts ($) | 17,650 (29,099) | 18,130 (29,302)

11. Other Pre Specified Outcome: Number of Readmissions
Time Frame: 30-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
readmissions | 0.39 (0.68) | 0.38 (0.73)

12. Other Pre Specified Outcome: Number of Readmissions
Time Frame: 90-day from indexed hospital discharge
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 389 | 393
readmissions | 0.92 (1.28) | 0.94 (1.41)

13. Other Pre Specified Outcome: Number of Readmissions
Description: Outcome is the number of hospital readmissions within 365-days from index hospital discharge and is reported for the subset of participants for which sufficient time has passed that 365-day outcomes can be observed in hospital claims data.
Time Frame: 365-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

14. Other Pre Specified Outcome: Any Hospital Use (Inpatient or ED)
Time Frame: 365-day from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

15. Other Pre Specified Outcome: Time to Readmission (Days)
Description: Outcome is the number of days until readmission for the subset of participants for which sufficient time has passed that 365-day outcomes can be observed in hospital claims data and who had a readmission within 365 days.
Time Frame: Up to 365 days from indexed hospital discharge
Reporting Status: Not Posted, anticipated posting 2021-01

16. Other Pre Specified Outcome: Number of Readmissions (for Patients With 3+ Readmissions in the Prior Year)
Time Frame: 180-day from indexed hospital discharge
Population: Pre-specified subset of patients with 3+ readmissions in the prior year who completed the 180-day primary outcome period.
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 224 | 222
readmissions | 1.95 (2.24) | 1.86 (2.12)

17. Other Pre Specified Outcome: Number of Readmissions (for Patients With 2 Readmissions in the Prior Year)
Time Frame: 180-day from indexed hospital discharge
Population: Pre-specified subset of patients with 2 readmissions in the prior year who completed the 180-day primary outcome period.
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 165 | 171
readmissions | 0.99 (1.38) | 1.09 (1.68)

18. Other Pre Specified Outcome: Number of Readmissions (for English Speaking Patients)
Time Frame: 180-day from indexed hospital discharge
Population: Pre-specified subset of English-speaking patients who completed the 180-day primary outcome period.
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 309 | 329
readmissions | 1.53 (1.85) | 1.53 (2.01)

19. Other Pre Specified Outcome: Number of Readmissions (for Non-English Speaking Patients)
Time Frame: 180-day from indexed hospital discharge
Population: Pre-specified subset of non-English speaking patients who completed the 180-day primary outcome period.
Measure: Mean (Standard Deviation); unit: readmissions
Arm/Group | Standard Care | Link2Care
Number analyzed (Participants) | 80 | 64
readmissions | 1.58 (2.44) | 1.48 (1.81)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 365 days post discharge from the index hospital admission. Because we measure outcomes through administrative records rather than clinical visits, records of adverse events also come from administrative records, such as the National Death Index. Some data are not yet available because of time lags from when events occur to when data is available to researchers. We report all known adverse events, with additional future data analysis planned.
Description: Serious adverse events are either death or the release of private health information (PHI) to parties external to the study team. Study targets high-risk population with expected mortality, unrelated to the study. Adverse Events are events that lead to readmission to the hospital for a study participant. The Camden Coalition conducted root-cause analysis to ascertain an AE's relatedness to the intervention, but had no contact with control group. AE are reported from hospital administrative data.
Arm/Group | Standard Care | Link2Care
All-Cause Mortality (participants affected / at risk) | 49/389 | 45/393
Serious Adverse Events (participants affected / at risk) | 0/389 | 0/393
Other Adverse Events (participants affected / at risk) | 240/389 | 245/393
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=389) | Link2Care (N=393)
Hospital Admission (Social circumstances) | 240 (599) | 245 (599) — Hospital admission (all causes/organ systems included here, as we are unable to track with this level of specificity).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Original RCT: Health Care Hotspotting Analysis Plan (2014-03-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT02090426/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Extension study: Medicaid outpatient outcomes (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT02090426/SAP_001.pdf